CLINICAL TRIAL: NCT05204511
Title: Exercise and Post-COVID/Long-COVID: Effects of Different Training Modalities on Physical Performance, Heart Rate Variability, Inflammation, Health-Related Quality of Life, Cognitive Function and Post-COVID/Long-COVID19 Symptoms
Brief Title: Exercise and Post-COVID/ Long-COVID: Effects of Different Training Modalities on Various Parameters in People Affected by the Sequelae of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel König, Principal Investigator, University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00726
Record Dates: First submitted 2022-01-21; First posted 2022-01-24 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Long COVID-19; Post-COVID-19 Syndrome; COVID-19
Keywords: exercise; exercise therapy; endurance training; concurrent training; physical peformance; inflammatory markers; quality of life; concentration performance; heart rate variability
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Motor Activity | interventions — Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post-COVID/Long-COVID endurance training group (Experimental): Participants affected by Post-COVID/Long-COVID that carry out a 12-week thrice weekly endurance training intervention
  Interventions: Other: endurance training
- Post-COVID/Long-COVID concurrent training group (Experimental): Participants affected by Post-COVID/Long-COVID that carry out a 12-week thrice weekly concurrent training intervention
  Interventions: Other: concurrent training
- Post-COVID/Long-COVID control group (No Intervention): Participants affected by Post-COVID/Long-COVID that don't carry out an exercise intervention

INTERVENTIONS:
Other: endurance training — endurance training of low to moderate intensity on a bicycle ergometer, crosstrainer or treadmill performed for 30-60 minutes per session
  Arms: Post-COVID/Long-COVID endurance training group
Other: concurrent training — combination of endurance training of low to moderate intensity on a bicycle ergometer, crosstrainer or treadmill performed for 20-40 minutes per session and resistance training of moderate intensity performing 2-3 sets of leg press, leg curls, chest press and seated horizontal rows
  Arms: Post-COVID/Long-COVID concurrent training group

SUMMARY:
The current COVID-19 pandemic is the most severe health crisis of the 21st century. This is not only due to the deaths caused by the disease. People that were affected by COVID-19 and supposedly recovered may suffer from long lasting sequelae. The presence of symptoms longer than 3 months after the infection with SARS-CoV-2 is referred to as Post-COVID-19 Syndrome or Long COVID-19. It is estimated that 10-20 percent of all infected people are affected. The most common symptoms include persistent fatigue, reduced physical capacity, dyspnoea, ageusia, anosmia, musculoskeletal pain and neuropsychological complaints such as depression, anxiety, insomnia and a loss of concentration.

Considering the novelty of the pathology, evidence on the successful treatment of Post-COVID/Long-COVID is scarce. Physical activity has been established as a treatment option for chronic diseases that have similar symptomatic manifestations to those of Post-COVID/Long-COVID. For example, exercise therapy has shown positive effects on the health status of patients with lung disease, depression, anxiety, insomnia and cognitive impairment. However, there has been controversy whether so-called Graded Exercise Therapy (GET) is a safe treatment strategy for patients with Chronic Fatigue Syndrome (CFS). This population may experience Post Exertional Malaise (PEM), a worsening of symptoms after physical, cognitive or emotional exertion. Since COVID-19 might be an infectious trigger for CFS, particular caution has to be taken when recruiting participants and when screening them for adverse events and worsening of symptoms during an exercise intervention.

It can be hypothesized that patients suffering from Post-COVID/Long-COVID can benefit from exercise in various ways, guaranteed that there is sufficient screening for PEM before and during the intervention and training volume and intensity are increased slowly and progressively.

The current study investigates the effects of two different training modalities, endurance training and a combination of endurance training and resistance training, on various parameters in people affected by Post-COVID/Long-COVID.

ELIGIBILITY:
Inclusion Criteria:

* laboratory-confirmed infection with SARS-CoV-2 via PCR a minimum of 12 weeks ago
* presence of at least one or more of persistent symptoms that can be attributed to Post-COVID/Long-COVID or a manifestation of reduced physical performance capacity since the infection with SARS-CoV-2

Exclusion Criteria:

* previous or current hospitalization due to the COVID-19 disease
* regular engagement in endurance or strength training (more than once per week) in the six months prior to enrollment
* contraindications for physical endurance and resistance exercise according to the guidelines of the American College of Sports Medicine (ACSM)
* clinical diagnosis of depression
* clinical diagnosis of anxiety
* clinical diagnosis of a sleep disorder
* clinical diagnosis of a cognitive deficit disorder
* a grade of 3 or higher on the Post-COVID-19 Functional Status Scale (PCFS)
* presence of post exertional malaise (PEM)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change of peak oxygen consumption (VO2peak measured in ml/min/kg) | Baseline - 6 weeks - 12 weeks
  VO2peak will be assessed during cardio pulmonary exercise testing (CPET) on a bicycle ergometer.

SECONDARY OUTCOMES:
Change of maximum lower body isometric muscle strength (measured in N) | Baseline - 6 weeks - 12 weeks
  Maximum lower body isometric muscle strength will be assessed via a leg press with integrated isometric force measurement (Compass 530, Suessmed GmbH).
Change of maximum hand grip strength (measured in kg) | Baseline - 6 weeks - 12 weeks
  Maximum hand grip strength will be assessed via a hand grip dynamometer (Saehan SH5001).
Change of Standard Deviation of RR-Intervals (SDNN measured in ms) | Baseline - 6 weeks - 12 weeks
  SDNN will be assessed via a short-term heart rate variability (HRV) measurement (BioSign).
Change of Root Mean Square of Successive Differences (RMSSD measured in ms) | Baseline - 6 weeks - 12 weeks
  RMSSD will be assessed via a respiratory sinus arrythmia measurement (BioSign).
Change of high-sensitive C-reactive protein (hs-CRP measured in mg/l) | Baseline - 6 weeks - 12 weeks
  hs-CRP will be assessed via blood sample.
Change of interleukin-6 (IL-6 measured in pg/ml) | Baseline - 6 weeks - 12 weeks
  IL-6 will be assessed via blood sample.
Change of tumor necrosis factor alpha (TNF-α measured in pg/ml) | Baseline - 6 weeks - 12 weeks
  TNF-α will be assessed via blood sample.
Change of health-related quality of life (HQoL) assessed via the SF-36 1.0 | Baseline - 6 weeks - 12 weeks
  The SF-36 1.0 is self-administered questionnaire and will be scored according to RAND (numeric value of 0-100). A high score represents a more favorable health status.
Change of mean time "correct rejection" (CR, speed during concentrated working measured in s) | Baseline - 6 weeks - 12 weeks
  CR will be assessed via Cognitrone (Schuhfried GmbH), which is a carefully administered computer test. Participants will be given the task of comparing a series of geometric figures.
Change of the number of present Post-COVID/Long-COVID specific symptoms | Baseline - 6 weeks - 12 weeks
  The number of Post-COVID/Long-COVID specific symptoms will be assessed using a list of symptoms provided by the National Institute for Health Care and Excellence (NICE). Each item will be referenced to as existent (yes) or non-existent (no) during the last 7 days.
Change of fatigue assessed via the Fatigue Severity Scale (FSS) | Baseline - 6 weeks - 12 weeks
  The FSS is a 9-item self-report questionnaire using a 1-7 Likert-scale
Change of dyspnoea assessed via the modified Medical Research Council (mMRC) dyspnoea scale | Baseline - 6 weeks - 12 weeks
  The mMRC dyspnoea scale measures perceived breathlessness and classifies subjects into dyspnoea grades from 0-4.
Change of absolute body fat (BF measured in kg) | Baseline - 6 weeks - 12 weeks
  BF will be assessed via a bioelectrical impedance analysis (seca BCA01A).
Change of absolute lean body mass (LBM measured in kg) | Baseline - 6 weeks - 12 weeks
  LBM will be assessed via a bioelectrical impedance analysis (seca BCA01A).
Change of step count per day | daily for 12 weeks starting with the first day of the intervention period
  Step count will be assessed daily during the 12-week intervention period using a wearable device (Polar Unite)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport Science, University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No